CLINICAL TRIAL: NCT04825639
Title: A Retrospective Study to Evaluate the Prevalence of Acute Kidney Injury in Patients With DKA and Sepsis
Brief Title: Identifying Risk Factors for Developing AKI in Sepsis
Status: Completed | Type: Observational
Sponsor: Cardiff and Vale University Health Board (Other Government)
Responsible Party: Sponsor
Other Study IDs: 20/DEC/8064
Record Dates: First submitted 2021-03-26; First posted 2021-04-01 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Sepsis; Acute Kidney Injury; Diabetic Ketoacidosis
MeSH Terms: conditions — Sepsis; Acute Kidney Injury; Diabetic Ketoacidosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sepsis: Patients admitted to PICU who are selected from registry based on primary diagnoses with codes for the following search codes were selected:
  Sepsis is defined as per the International Consensus Conference pediatric sepsis definition (2005) [citation 1].
  In silico analysis will be carried out in the sepsis cohort comparing admissions with Acute Kidney Injury (AKI) and those without AKI to identify factors associated with AKI.
  In those selected admissions to PICU, information on Renal Function, Chloride levels, clinical outcome and medication use as well as fluid resuscitation will be collected from hospital online resources such as discharge summaries, results portal and the PICANet database. In addition the Paediatric Index of Mortality 3 severity of illness scores will be reported for all admissions.
  Sepsis will be defined based on the International Pediatric Consensus Conference definition of sepsis (2005)
  Interventions: Other: No intervention
- Diabetic Ketoacidosis (DKA): This group is defined based on the British Society of Paediatric Endocrinology and Diabetes.case definition for Diabetic Ketoacidosis [citation 2].
  The data collected will be similar to the sepsis cohort. In silico analysis will be carried comparing those with AKI and without AKI in the DKA cohort.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — no intervention

SUMMARY:
A study to evaluate the prevalence of Acute Kidney Injury (AKI) in patients with Diabetic Ketoacidosis (DKA) and sepsis using data collected prospectively to a patient registry. The primary objective is to compare the prevalence of AKI in sepsis and DKA in different age groups in children and investigate the difference in the prevalence of hyperchloremia in the two groups.Secondary objectives are Compare the prevalence of AKI in sepsis and DKA in different age groups in children and investigate the difference in the prevalence of hyperchloremia in the two groups.

DETAILED DESCRIPTION:
It is a descriptive study to report the prevalence ofAcute Kidney Injury ( AKI) in the two cohorts of sepsis and Diabetic Ketoacidosis ( DKA). In addition we aim to evaluate the relation with hyperchloremia. In both groups, attempts will be made to evaluate the association of risk factors such as severity of dehydration/shock and hyperchloremia with AKI in the two groups.

Data will be analysed using SPSS software. Categorical variables will be analysed using Chi-square test and if appropriate, multiple logistic regression analysis. Continuous variable will be analysed with Student's T test and if possible, by linear regression modelling. The differences between the two groups may analysed using Analysis of Variance (ANOVA).

The study will collect anonymous data from 2015 to 2020 from the Paediatric Intensive Care Audit Network (PICANet) database for a tertiary PICU servicing the pediatric population of Wales.This data is submitted prospectively for audit of clinical outcomes of children admitted for paediatric intensive care in the United Kingdom. The study was reviewed by the Institutional Research and Development department and was given exemption for ethics committee review as it does not involve direct patient contact and the data is anonymous. Approval was obtained from the relevant database manager, institutional information governance department as well as the Health Care Research Wales.

ELIGIBILITY:
Inclusion Criteria

* Children under 16 years and admitted to PCCU or wards in the past 5 years
* Diagnosis of DKA or Sepsis/severe bacterial infection/septic shock

DKA - defined as per the British Society for Paediatric Endocrinology and Diabetes (BSPED) guidance. Sepsis is defined based on the International Pediatric Sepsis Consensus Conference guidance (2005)

8.3. Exclusion Criteria

* Any patients identified as above but not able to obtain case notes for any reason.
* Patients with pre-existing kidney conditions
* Patients with inborn errors of metabolism

Ages: 0 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Study Population: Children admitted to PICU with sepsis as per the sepsis consensus conference (2005) definition.
  Children with DKA admitted to PICU and wards. Diabetic Ketoacidosis defined based on the British Paediatric Society of Endocrinology and Diabetes.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of Acute Kidney Injury in the sepsis and DKA cohorts | during admission to PICU
  Acute Kidney Injury will be defined based on the Kidney Disease Improving Global Outcomes (KDIGO) 2012 [citation 3] guidelines. Serum Creatinine and Urine output will be used for defining Acute Kidney Injury. Serum creatinine is measured in microMol/litre and urine output in millilitres (ml)

SECONDARY OUTCOMES:
Risk factors associated with AKI | During admission to PICU
  Various risk factors will be evaluated such as cardiac arrest prior to admission or during admission, mechanical ventilation, hypotension or shock requiring vaso-active medications as well as use of medications which may be nephrotoxic.
Compare chloride levels in the AKI and non AKI groups | during admission in PICU
  The units used for Chloride levels is mMol/Litre

CONTACTS AND LOCATIONS:
Locations (1):
- Noah's Ark Children's hospital, Cardiff, South Glamorgan, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 2. Link to the guidelines documents accessed on 29/03/3-21:https://www.bsped.org.uk/media/1798/bsped-dka-guideline-2020.pdf
- [Background] Kidney Disease: Improving Global Outcomes (KDIGO) clinical practice guideline for acute kidney injury.Kidney Int Suppl. 2012;2:1-141. doi: 10.1038/kisup.2012.3
- [Result] Goldstein B, Giroir B, Randolph A; International Consensus Conference on Pediatric Sepsis. International pediatric sepsis consensus conference: definitions for sepsis and organ dysfunction in pediatrics. Pediatr Crit Care Med. 2005 Jan;6(1):2-8. doi: 10.1097/01.PCC.0000149131.72248.E6. PMID 15636651